CLINICAL TRIAL: NCT07102160
Title: A Prospective, Multi-Center, Open-Label Clinical Investigation of the Cleaner Vac® Thrombectomy System for Treatment of Lower Extremity Proximal Deep Vein Thrombosis (DVT)
Brief Title: Cleaner Long-tErm Assessment Registry - Venous Insights and Efficacy With eXtended Tracking
Acronym: CLEAR-VIEW XT
Status: Recruiting | Type: Observational
Sponsor: Argon Medical Devices (Industry)
Collaborators: Avania (Industry); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CNPV01
Record Dates: First submitted 2025-07-11; First posted 2025-08-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Deep Vein Thrombosis (DVT); Thrombus in the Peripheral Venous Vasculature; Venous Embolism; Thrombus in the Central and Peripheral Circulatory System, Including Saphenous Vein Grafts
Keywords: Aspiration Thrombectomy; Deep Vein Thrombosis (DVT); Peripheral VTE; Venous thromboembolism; Percutaneous mechanical thrombectomy
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- DVT Subgroup: This is a defined cohort focused on patients with lower extremity proximal deep vein thrombosis (DVT) who will undergo treatment with Cleaner Vac® Thrombectomy System. Participants will complete required follow-up at discharge and at 1, 6, 12, and 24 months.
  Interventions: Device: Aspiration thrombectomy system

INTERVENTIONS:
Device: Aspiration thrombectomy system — The Cleaner Vac® Thrombectomy System is a percutaneous mechanical aspiration thrombectomy device designed for the removal of fresh, soft thrombi and emboli from the peripheral venous vasculature. The system includes an aspiration canister with integrated pump, an 18F aspiration catheter, a handpiece with aspiration control lever, a dilator, and an optional flushing adapter. The device operates via controlled suction to extract thrombus and restore venous patency.

SUMMARY:
The primary objective of this clinical investigation is to evaluate the safety and effectiveness of the Cleaner Vac® Thrombectomy System for the treatment of thrombus in patients with lower extremity proximal deep vein thrombosis (DVT). This prospective, multi-center, open-label study will assess clinical outcomes, device performance, and procedural success in a single DVT study cohort.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for the study:

1. At least 18 years of age at the time of consent.
2. Undergo frontline (primary) treatment with Cleaner Vac® Thrombectomy System in the peripheral venous vasculature and have at least one component introduced into the body.
3. Written informed consent obtained through the IRB-approved ICF.

   For the DVT cohort, participants must meet all criteria above and below to be eligible for the study:
4. Present with unilateral or bilateral lower extremity DVT involving at least one of the following veins:

   1. Femoral-popliteal vein
   2. Common femoral vein
   3. Iliac vein
   4. Inferior Vena Cava (IVC)
5. DVT diagnosis confirmed by imaging within 14 days of the index procedure.
6. Symptomatic DVT with onset within 6 weeks of enrollment.

Exclusion Criteria:

Subjects will be excluded from the study if any of the following criteria are met:

1. Contraindication to systemic or therapeutic doses of anticoagulants.
2. Contraindication to iodinated contrast that cannot be adequately premedicated.
3. Life expectancy less than 1 year due to advanced malignancy, as determined by the investigator at the time of enrollment
4. Patients that are pregnant.
5. Known coagulation disorders both acquired (Heparin Induced Thrombocytopenia, etc.) or genetic (e.g., Factor V Leiden, etc.), thrombophilia, or hypercoagulable states that, in the opinion of the Investigator, cannot be medically managed throughout the study period.
6. Treatment of target venous segment with thrombolytics within previous 14 days of the index procedure.
7. Known congenital anatomic anomalies of the inferior vena cava (IVC) or iliac veins.
8. Known history of a Patent Foramen Ovale (PFO).
9. Hemoglobin < 8.0 g/dL, INR > 2.0 before warfarin was started, or platelets < 50,000/µl which cannot be corrected prior to enrollment.
10. Severe renal impairment (estimated GFR < 30 ml/min) in patients who are not yet on dialysis. Patients with GFR <30 ml/min who are already on dialysis can be enrolled.
11. Patients with intermediate-high risk or high-risk pulmonary embolism (PE) defined as follows:

    1. High-risk PE: Presence of hemodynamic instability, including cardiac arrest, obstructive shock (systolic blood pressure <90 mmHg or need for vasopressors with signs of end-organ hypoperfusion), or persistent hypotension (systolic BP <90 mmHg or a drop ≥40 mmHg for >15 minutes not due to other causes)
    2. Intermediate-high-risk PE: Hemodynamically stable patients with both right ventricular (RV) dysfunction (on echocardiography or CT) and elevated cardiac biomarkers (e.g., troponin).
12. Complete infrarenal IVC occlusion.
13. Chronic non-ambulatory status.
14. Current enrollment in another investigational device or drug study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 185 adult participants undergoing percutaneous mechanical thrombectomy using the Cleaner Vac® Thrombectomy System for the treatment of thrombus in the peripheral venous vasculature.
  Participants must be at least 18 years old and undergoing frontline treatment with the Cleaner Vac® device. The DVT subgroup must have symptomatic, imaging-confirmed DVT involving the femoral-popliteal, common femoral, iliac veins, or inferior vena cava (IVC), with symptom onset within 6 weeks and imaging confirmation within 14 days of the index procedure.
  The study population is intended to reflect a real-world, all-comers cohort treated across up to 50 investigational sites in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Technical Success | At the time of the index procedure
  ≥75% thrombus removal in the target venous segment, assessed by change in Marder Score
Composite rate of Major Adverse Events (MAEs) within 30 days post-procedure | 30 days post-index procedure

SECONDARY OUTCOMES:
Freedom from Device- or Procedure-Related Serious Adverse Events (SAEs) | 30 days post-procedure
Post-Thrombotic Syndrome Severity | Up to 24 months
  Assessment of post-thrombotic syndrome using the Villalta score, which combines patient-reported symptoms and clinician-assessed signs to generate a composite score. A score ≥5 indicates the presence of post-thrombotic syndrome, with higher scores reflecting greater severity.
Venous patency | From 30 days post-treatment to the end of the study period
  Presence of flow in the treated venous segment without re-thrombosis
Need for Target Vessel Reintervention | From date of index procedure up to 24 months
  Any additional endovascular or surgical procedure to address recurrent/residual thrombus
Numeric Pain Rating Scale | Up to 24 months
  Self-reported health status measured using the Numeric Pain Rating Scale questionnaire, which evaluates current, best, and worst pain experienced on a 0 (minimum) to 10 (maximum) level scale. 10 having worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Danyel Carr, MS, Study Director — Argon Medical Devices; Pete Stibbs, MD, MSc, MBA, Study Director — Argon Medical Devices
Locations (3):
- United States (3):
  - Baycare Health System, Tampa, Florida
  - St. Elizabeth Healthcare - Edgewood, Edgewood, Kentucky
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Argon Medical Devices - CLEAR-VIEW XT study information — https://www.argonmedical.com/research/cleaner-long-term-assessment-registry/